CLINICAL TRIAL: NCT06293911
Title: Clinical Comparison of a Postbiotic-gel With Placebo Gel for Gingival Inflammation in Patients With Down Syndrome: Randomized Clinical Trial
Brief Title: Clinical Comparison of a Postbiotic-gel With Placebo Gel for Gingival Inflammation in Patients With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-POSTBIOTICSDOWNSYNDROME
Record Dates: First submitted 2024-02-25; First posted 2024-03-05 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Down Syndrome; Gingival Bleeding
MeSH Terms: conditions — Down Syndrome; Gingival Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postbiotic group (Experimental)
  Interventions: Other: Biorepair Plus Parodontgel Intensive
- Placebo group (Active Comparator)
  Interventions: Other: Placebo gel

INTERVENTIONS:
Other: Biorepair Plus Parodontgel Intensive — The Biorepair Plus Parodontgel Intensive gel will be used after home oral hygiene once a day.
  Arms: Postbiotic group
Other: Placebo gel — The placebo gel (without hyaluronic acid, Lactobacillus Ferment, Aloe Barbadensis Leaf Juice Powder and lactoferrin) will be used after home oral hygiene once a day.
  Arms: Placebo group

SUMMARY:
The aim of the study is to evaluate the efficacy of home treatment with a postbiotic-based gel for the management of periodontal inflammation in patients with Down syndrome.

Patients will be enrolled at the S.C. Odontostomatologia dell'Azienda Ospedaliera "Ordine Mauriziano di Torino", Turin, Italy. After the collection of the periodontal clinical indexes (BoP%, PCR%, dental mobility, mMGI, compliance and satisfaction questionnaire), patients will undergo a professional mechanical debridement with ultrasonic instruments and glycine powders.

Then, they will be randomly divided into two groups according to the home treatment:

* in the Trial group Biorepair Plus Parodontgel Intensive (containing microRepair®, hyaluronic acid, Lactobacillus Ferment and Aloe Barbadensis Leaf Juice Powder) will be used once a day for all the duration of the study
* in the Control group, a placebo gel without (active ingredients) will be used once a day for all the duration of the study.

Indexes will be re-evaluated after 1 (T1), 3 (T2) and 6 months. The professional mechanical debridement will be performed again at T3 timepoint.

ELIGIBILITY:
Inclusion Criteria:

* not bedridden patients with Down syndrome
* gingival inflammation and bleeding

Exclusion Criteria:

* lack of compliance signalled by caregivers
* other systemic diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Change in Bleeding on Probing (BOP%) | Baseline (T0), after 1 month (T1), 3 months (T2) and after 6 months (T3)
  Dichotomous scoring (yes/no) of bleeding sites on 4 surfaces of teeth.
Change in Plaque Control Record (PCR%) | Baseline (T0), after 1 month (T1), 3 months (T2) and after 6 months (T3)
  % assessment of the amount of plaque on dental surfaces; it is detected on 4 surfaces: distal, mesial, vestibular, lingual / palatal. The number of sites with plaque is divided by the total number of sites available in the mouth and multiplied by 100. Results indicate the index as a percentage.
Change in Dental mobility | Baseline (T0), after 1 month (T1), 3 months (T2) and after 6 months (T3)
  Scoring criteria
  Grade 0: oscillation within 0.2 mm; the teeth move naturally and there are no mobility problems; Grade I: horizontal mobility of the tooth from 0.2 to 1 mm; Grade II: horizontal mobility of the tooth from 1 to 2 mm; Grado III: horizontal mobility equal to or greater than 3 mm or vertical mobility of the tooth.
Change in Modified Gingival Index | Baseline (T0), after 1 month (T1), 3 months (T2) and after 6 months (T3)
  Scoring criteria (one measurement for each tooth: upper first incisors, first premolars/first primary molars and first molars):
  0. Absence of inflammation
  Mild inflammation (marginal or papillary unit) Mild inflammation (entire marginal and papillary unit) Moderate inflammation Severe inflammation
Change in compliance | Baseline (T0), after 1 month (T1), 3 months (T2) and after 6 months (T3)
  Subjective evaluation of the patient's degree of compliance with the proposed treatment by Visual Analogue Scale (VAS), assessing compliance with dosage, alterations and modifications on lifestyle, and adherence to set recalls; to which is associated a score from 0 to 10 of which:
  * 0 to 2: Poor compliance;
  * 3 to 5: Sufficient compliance;
  * 6 to 8: Good compliance;
  * 9 to 10: Excellent compliance.
Change in product satisfaction | Baseline (T0), after 1 month (T1), 3 months (T2) and after 6 months (T3)
  * Product liking questionnaire: evaluation of taste, smell, consistency, persistence and ease of application by Visual Analogue Scale (VAS) and filling out a questionnaire to which a score from 0 to 10 is associated, of which:
  * 0: Insufficient;
  * 1 to 3: Sufficient;
  * 4 to 6: Good;
  * 7 to 9: Very Good;
  * 10: Excellent.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD, Principal Investigator — University of Pavia
Locations (1):
- S.C. Odontostomatologia - Azienda Ospedaliera "Ordine Mauriziano di Torino", Turin, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to the Principal Investigator.